CLINICAL TRIAL: NCT00399373
Title: Structuring the Integration of Services For Medicaid Recipients With Chronic Illness, Substance Abuse Problems and Possible Psychiatric Disorders
Brief Title: Structuring the Integration of Care Management Services For Medicaid Enrollees Recipients With Chronic Illness, Substance Abuse Problems and Possible Psychiatric Disorders
Status: Terminated | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00001352; 100326 (CHCS)
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Chronic Illness
Keywords: disease management; substance abuse
MeSH Terms: conditions — Chronic Disease; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Quality Improvement Initiative: The initial step in the quality improvement initiative was a letter sent from JHHC Care Management Department to the quality improvement initiative group, inviting them to take advantage of the case management services that are part of their current benefits in the Priority Partners MCO. It is similar to the standard letter sent to PPMCO members who are appropriate for a JHHC disease or case management program. A substance abuse outreach staff initiated telephonic contact with the members in the intervention group. The staff member then refered to substance abuse treatment when possible and appropriate and refered to medical case management.
- Control group: No additional improvement modalities

SUMMARY:
The study seeks to measure the effect of increased coordination of care on medical costs, treatment utilization and selected clinical indicators among a Medicaid population with chronic medical conditions and substance abuse problems? We shall address this question by conducting a demonstration project consisting of the provision of integrated care management (somatic and behavioral) to Medicaid enrollees living on the Eastern Shore of Maryland and who have both chronic medical conditions and problems with substance abuse. A specific component of the study will be the participation of Maryland's Mental Health Administration (MHA) and MAPS, the administrator of psychiatric services for the Medicaid enrollees in Maryland. We shall compare the results of the integrated care management for the study sample on the Eastern Shore with a control group from the counties of western Maryland.

DETAILED DESCRIPTION:
Problem in context. In an environment of increased competition for governmental funding, Medicaid programs in every state are bracing for decreased resources being available for the care of their enrollees. A possible result of less funding is reduced quality of healthcare. In response to this threat, The Center for Health Care Strategies, Inc, (CHCS) a non-profit organization dedicated to improving the quality of publicly financed health care, issued an RFP for participation in a multisite project to expand or enhance existing efforts to improve the way care for Medicaid enrollees with multiple chronic conditions is delivered, integrated, measured and financed.

Present knowledge. While there is strong documentation of improved population health status with care management, the evidence for the immediate economic effects of care management initiatives is mixed for commercial and absent for Medicaid populations. CHCS is presently conducting a multisite study (in which we participate) of whether or not a business case (return on investment) can be made for quality improvement initiatives in a Medicaid population.

Research question. What is the effect of increased coordination of care on medical costs, treatment utilization and selected clinical indicators among a Medicaid population with chronic medical conditions and substance abuse problems? We shall address this question by conducting a demonstration project consisting of the provision of integrated care management (somatic and behavioral) to Medicaid enrollees living on the Eastern Shore of Maryland and who have both chronic medical conditions and problems with substance abuse. A specific component of the study will be the participation of Maryland's Mental Health Administration (MHA) and MAPS, the administrator of psychiatric services for the Medicaid enrollees in Maryland. We shall compare the results of the integrated care management for the study sample on the Eastern Shore with a control group from the counties of western Maryland.

The primary goal of the project will be to improve the coordination of medical, substance abuse and mental health services for a group of Medicaid beneficiaries with chronic medical conditions. We hypothesize that the recipients of integrated care management (on the Eastern Shore) will have lower total medical costs (pharmacy, inpatient and outpatient), higher utilization of mental health and substance abuse services and lower use of emergency department services than those who received customary care (in western Maryland).

The secondary goal of this project will be to assist in the further development and piloting of information systems within MHA that will facilitate sharing of clinical information necessary for the coordination of behavioral (mental health and substance abuse) and medical care management between a Medicaid MCO (JHHC's PPMCO) and the mental health carve-out ASO, MAPS-MD. The outcome measurement for the secondary objective will be the extent to which an information system for coordination of care and population based queries has been established within MHA and is, with proper oversight by MHA, accessible to responsible entities.

Significance. The project targets a vulnerable population within Medicaid enrollees that are challenged when accessing care and are responsible for high total medical costs. The results of the project should be helpful to other the MCOs in Maryland's Health Partners, as well as to states with similar Medicaid systems as they seek to provide integrated healthcare services to their populations.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years of age or older;
2. Resident of one of the following Maryland counties: Caroline, Cecil, Kent, Queen Anne's, Talbot, Dorchester, Somerset, Wicomico, Worcester, Allegheny, Frederick, Garrett, Washington, Calvert, Charles, or St. Mary's; or
3. Chronic medical condition(s) identified by ACG Case Mix software (e.g. an ACG score => 0.10) as likely to incur high costs in the following year; and
4. Substance use problem in the past 27 months as indicated by an ICD-9 code or CPT code on DHMH list for Special Needs Population.

Exclusion Criterion.

1) Enrolled in or eligible for enrollment in a Special Needs disease management program at JHHC: HIV/AIDS, Partners with Mom, Omega Life. It is necessary to exclude these programs because PPMCO members are already receiving intensive care management.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We determined the size of the quality improvement initiative sample by the case management resources available at JHHC. Without adding personnel, the maximum number of new cases that can be assumed by the 3.5 (FTE) JHHC case managers for the Eastern Shore is 130.
Sampling Method: Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2005-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Total medical costs (per member per month) | monthly average, calculated at the end of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Fagan, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins HealthCare LLC, Glen Burnie, Maryland, United States